CLINICAL TRIAL: NCT01616784
Title: The Relative Effectiveness of Pumps Over Multiple Dose Injections and Structured Education Trial
Brief Title: The REPOSE (Relative Effectiveness of Pumps Over MDI and Structured Education) Trial
Acronym: REPOSE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: Cambridge University Hospitals NHS Foundation Trust (Other); NHS Dumfries & Galloway (Other); NHS Lothian (Other Government); NHS Greater Glasgow and Clyde (Other); Harrogate & District NHS Foundation Trust (Other); King's College Hospital NHS Trust (Other); Nottingham University Hospitals NHS Trust (Other); National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH15295; 08/107/01 (Other Grant/Funding Number: HTA); 2010-023198-21 (EudraCT Number); 11/H1002/10 (Registry Identifier: REC); 61215213 (Registry Identifier: ISRCTN); 10997 (DRN 628) (Registry Identifier: UKCRN)
Record Dates: First submitted 2012-05-02; First posted 2012-06-12 (Estimated); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Type 1 Diabetes
Keywords: Adult; Diabetes Mellitus; Type 1; Humans; Hypoglycemic Agents; Administration and Dosage; Insulin; Self Care; Health Education; Insulin Infusion Systems; Randomised controlled trial; Patient Education as Topic; Hemoglobin A; Glycosylated
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance; Health Education | interventions — Insulin Detemir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Multiple daily injections plus DAFNE (Active Comparator): Optimised MDI therapy using rapid and twice daily (Detemir/Levemir) long-acting insulin analogues
  Interventions: Other: MDI (levemir® & quick acting insulin) plus DAFNE
- CSII (Insulin Pump) plus DAFNE (Experimental): Medtronic MiniMed Paradigm Veo Insulin pumps (X54)
  Interventions: Other: CSII (Insulin Pump) plus DAFNE

INTERVENTIONS:
Other: CSII (Insulin Pump) plus DAFNE — Medtronic MiniMed Paradigm Veo Insulin pumps (X54)
  Other Names: Continuous subcutaneous insulin infusion; CSII; external insulin pumps
  Arms: CSII (Insulin Pump) plus DAFNE
Other: MDI (levemir® & quick acting insulin) plus DAFNE — Optimised MDI therapy using rapid and twice daily (Detemir/Levemir) long-acting insulin analogues
  Arms: Multiple daily injections plus DAFNE

SUMMARY:
For type-1 diabetes, the aim of insulin therapy is to keep blood glucose close to normal while avoiding hypoglycaemia but this is severely limited by the relative crudeness of current insulin delivery in comparison with the physiology of the β-cells which secrete insulin. Insulin is generally administered by multiple injections MDI with the dose adjusted according to eating and exercise. Insulin can now also be administered using a pump (CSII), which is a device, roughly the size of a mobile phone and containing sufficient insulin to supply both the needs of basal metabolism throughout the day, and the boluses which have to cover meals. The use of CSII is expensive compared to injections, but there are important potential benefits which include improved glycaemic control, reduced risk of hypoglycaemia (low blood sugar) and a more flexible lifestyle and better quality of life. There have been no trials in adults that have compared CSII treatment with MDI where the same structured training in intensive insulin therapy has been given, so the precise benefit of the pump technology is still unclear. There is a need to establish this, and identify patients who benefit the most so that the Department of Health can calculate the proportion of adults that would benefit from CSII therapy and so ensure that commissioning bodies provide the necessary reimbursement. The aim of the trial is therefore to establish the added benefit of CSII therapy over multiple injections on glycaemic control and hypoglycaemia in individuals with Type 1 diabetes receiving similar high quality structured training (Dose Adjustment For Normal Eating:DAFNE) in insulin therapy. Additional assessments will include effects on quality of life and cost effectiveness.

DETAILED DESCRIPTION:
The trial is a multi-centre randomised controlled trial whereby between 40 and 49 type-1 diabetic, adult volunteers, aged 18 and above, will be recruited per site from 7 secondary care centres (Sheffield, Kings College Hospital London, Harrogate District Hospital, Addenbrookes Hospital Cambridge, Glasgow Royal Infirmary, Dumfries and Galloway Royal Infirmary and Edinburgh Royal Infirmary). The sites will be required to recruit participants to at least 3 CSII DAFNE (Dose Adjustment for Normal Eating)courses and 3 MDI DAFNE courses. This will mean that in total on the trial, 140 participants are randomised to CSII and 140 to MDI. Participants will be recruited through direct approach if already on the waiting list for a DAFNE course or through advertisement in various clinics.

ELIGIBILITY:
Inclusion Criteria:

* Is aged 18 yrs and above.
* Have had type-1 diabetes for at least 12 months (as assessed by date clinically diagnosed).
* Is fluent in speaking, reading and understanding English.
* Has no preference to either CSII or MDI arm of the study and is happy to be randomised.
* Is currently using or willing to switch to Detemir.
* Is willing to undertake self-monitoring of blood glucose (SMBG), carbohydrate counting and insulin self-adjustment. (Enrolment staff should check that any participant with a baseline HbA1c of above 12% is willing to complete SMBG).
* Has a need for structured education to optimise diabetes control in the opinion of the investigator.

Exclusion criteria:

* Inability to give informed consent.
* Is pregnant or planning to become pregnant within the next 2 years.
* Has used CSII within the last 3 years.
* Has already completed a diabetes education course.
* Has severe needle phobia.
* Has a current history of alcohol or drug abuse.
* Has a history of heart disease within the past 3 months.
* Has hypertension that is not under control with hypertensive medication (diastolic blood pressure >100mmHg and or sustained systolic level >160).
* Has renal impairment with a chance of needing renal replacement therapy within the next 2 years (Enrolment staff should check that creatinine levels are not above 200 µmol/L).
* Has recurrent episodes of skin infections.
* Has serious or unstable medical or psychological conditions.
* Has taken part in any other investigational clinical trial during the 4 months prior to screening.
* Has any other issue that may preclude the participant from satisfactory participation in the study based on investigatory judgement.
* Has a strong need for pump therapy in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2011-11; Primary Completion 2015-06 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The change in HbA1c after 2 years in those participants whose baseline HbA1c was at or above 7.5% (58mmol/mol). | 2 years
  The change in HbA1c after 2 years in those participants whose baseline HbA1c was at or above 7.5% (58mmol/mol).
  (Change will be calculated from baseline at 24 months)

SECONDARY OUTCOMES:
The proportion of participants reaching the NICE target of an HbA1c level of 7.5% (58mmol/mol) or less | 6, 12 and 24 months
  HbA1c is a measurement of glycosylated haemoglobin which reflects overall blood glucose values over the previous 6-8 weeks(24). This is regarded as the gold standard measure of glycaemic control. There is a strong relationship between HbA1c and the risk of developing long term diabetic complications and it is accepted as a surrogate for long term outcomes in individuals with diabetes.
  Since HbA1c can be measured by different techniques we will ensure standardisation by measuring HbA1c in blood samples at a central laboratory.
  (Change will be calculated from baseline at 24 months)
Diabetes specific quality of life | 6, 12 and 24 months
  DSQOL Diabetes-specific quality of life (QoL) will be assessed using the scale DSQOL.
  (Change will be calculated from baseline at 24 months)
Hypoglycaemia (severe & moderate) | 6, 12 and 24 months
  The investigators will record both severe and moderate episodes of hypoglycaemia in participants. This should increase power and identify the ability of CSII to reduce rates of hypoglycaemia. It will also be possible to assess the effects of both, by comparing quality of life measures in those with only moderate hypos, versus those with moderate and severe.
  (Change will be calculated from baseline at 24 months)
Insulin dose | 6, 12 and 24 months
  Some studies have indicated that CSII results in the use of less insulin. We will therefore record participants' self-reported insulin dose at each time point and calculate units/kg body weight.
  (Change will be calculated from baseline at 24 months)
Body weight | 6, 12 and 24 months
  If CSII treatment results in the use of less insulin, it may have a favourable effect on weight since with less insulin there is a propensity for the body to store fewer nutrients. We will therefore record weight at each time point of the trial.
  (Change will be calculated from baseline at 24 months)
Blood lipids & proteinuria | 6, 12 and 24 months
  Blood samples will be taken using local labs and lipids (including HDL cholesterol). Albumin- creatinine ratio (a sensitive measure of proteinuria) will be measured from urine samples.
  (Change will be calculated from baseline at 24 months)
Diabetic Ketoacidosis | 6, 12 and 24 months
  This outcome will be measured through the assessment of any SAE's and AEs.
  (Change will be calculated from baseline at 24 months)
Fear of hypoglycaemia | 6, 12 and 24 months
  The Hypoglycaemia Fear Scale (HFS) is a well validated psychometric tool assessing participants fear of hypoglycaemia both overall and in terms of behaviour and worry. It has been used to assess the impacts of different hypoglycaemic events such as severe, moderate and mild hypoglycaemic episodes on fear of hypoglycaemia (33). A specific benefit to the HFS is that it may be able to identify participants who are likely to maintain high blood glucose levels, thus aiding understanding of potential reasons for poor glycaemic control.
  (Change will be calculated from baseline at 24 months)
Diabetes Treatment Satisfaction | 6, 12 and 24 months
  The Diabetes Treatment Satisfaction Questionnaire (DTSQ measures treatment satisfaction which refers to an individual's subjective appraisal of their experience of treatment, including ease of use, side effects and efficacy. Improvements in satisfaction are not necessarily accompanied by improvements in QoL; treatment satisfaction can be high despite diabetes having a negative impact on QoL, which is why it is important to measure both separately.
  (Change will be calculated from baseline at 24 months)
Emotional Wellbeing | 6, 12 and 24 months
  The Hospital Anxiety and Depression Scale (HADS) measures anxiety on one subscale and depression on another through the use of 7 questions for each characteristic. It is important to measure emotional wellbeing in the trial as participants may find it easier to manage their condition after DAFNE education or with one of the treatments. This might have a substantial effect on their emotional wellbeing that the QoL measures are not sensitive enough to pick up.
  (Change will be calculated from baseline at 24 months)
Participant views regarding the pump/multiple injection course & treatment | 6, 12 and 24 months
  Participant post course interviews
  Participants will be interviewed regarding:
  1. Understandings of the trial and motivation for participation.
  2. Views about outcome of randomisation.
  3. Expectations/concerns about trial participation and (if relevant) change to CSII.
  4. Experience of/views about the course and (if relevant) change to CSII.
  5. Changes they have made to diabetes management since the course and short/long terms goals set.
  6. Likes/dislikes of CSII or MDI treatment. (Change will be calculated from baseline at 24 months)
Educator views regarding the pump/multiple injection course & treatment | 6, 12 and 24 months
  Educator post course interviews
  Educators will be interviewed regarding:
  a) Insight and experience of what took place on the course. b) Recommendations for future course development.
  c) Recommendations for support that should be offered to patients who move onto pumps.
  (Change will be calculated from baseline at 24 months)
Costs and Outcomes | 6, 12 and 24 months
  Costs and quality adjusted life years will be estimated for each individual recruited to the trial. Mean values for each arm will be calculated.
  (Change will be calculated from baseline at 24 months)
Incremental cost-effectiveness ratio | 6, 12 and 24 months
  Cost-effectiveness will be described using plots of incremental costs and QALYs on the cost-effectiveness plane, together with their associated cost-effectiveness acceptability curves and frontiers. The incremental cost-effectiveness ratio and the probability that CSII will be cost-effective in the range of £20,000-£30,000 per QALY will be the main focus.
  (Change will be calculated from baseline at 24 months)
Costs | 6, 12 and 24 months
  Mean values of cost wll be estimated and the value will be calculated for each individual
  (Change will be calculated from baseline at 24 months)
General Quality of Life | 6, 12 and 24 months
  This will be measured by 3 different measures, the WHOQOL bref, SF12 and EQ5D.
  (Change will be calculated from baseline at 24 months)
Quality of adjusted life years | 6, 12 and 24 months
  Mean values will be estimated and value will be calculated for each individual (Change will be calculated from baseline at 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Simon Heller, Prof, Principal Investigator — University of Sheffield
Locations (8):
- United Kingdom (8):
  - Addenbrookes Wolfson Diabetes and Endocrine Clinic, Box 281, Addenbrookes Hospital, Hills Road, Cambridge, Cambridgeshire
  - Harrogate District Hospital, Diabetes Centre, Lancaster Park Road,, Harrogate, North Yorkshire
  - Dumfries and Galloway Royal Infirmary, Diabetes Centre, Cluden West, Crichton Hall,, Dumfries, Scotland
  - Royal Infirmary of Edinburgh, Department of Diabetes, 51 Little France Crescent, Edinburgh, Scotland
  - Stobhill ACH, Diabetes Clinic, 133 Balornock Road, Glasgow, Scotland
  - Sheffield Teaching Hospital, Diabetes Centre, Northern General Hospital, PO Box 1, Herries Road, Sheffield, South Yorkshire
  - Kings College Hospital, Diabetes Centre, Suite 3, Golden Jubilee Wing, Denmark Hill, London
  - Nottingham University Hospitals NHS Trust, Queens Medical Centre Campus, Derby Road, Nottingham

REFERENCES:
- [Result] REPOSE Study Group. Relative effectiveness of insulin pump treatment over multiple daily injections and structured education during flexible intensive insulin treatment for type 1 diabetes: cluster randomised trial (REPOSE). BMJ. 2017 Mar 30;356:j1285. doi: 10.1136/bmj.j1285. PMID 28360027
- [Result] Heller S, White D, Lee E, Lawton J, Pollard D, Waugh N, Amiel S, Barnard K, Beckwith A, Brennan A, Campbell M, Cooper C, Dimairo M, Dixon S, Elliott J, Evans M, Green F, Hackney G, Hammond P, Hallowell N, Jaap A, Kennon B, Kirkham J, Lindsay R, Mansell P, Papaioannou D, Rankin D, Royle P, Smithson WH, Taylor C. A cluster randomised trial, cost-effectiveness analysis and psychosocial evaluation of insulin pump therapy compared with multiple injections during flexible intensive insulin therapy for type 1 diabetes: the REPOSE Trial. Health Technol Assess. 2017 Apr;21(20):1-278. doi: 10.3310/hta21200. PMID 28440211
- [Derived] Bradburn MJ, Lee EC, White DA, Hind D, Waugh NR, Cooke DD, Hopkins D, Mansell P, Heller SR. Treatment effects may remain the same even when trial participants differed from the target population. J Clin Epidemiol. 2020 Aug;124:126-138. doi: 10.1016/j.jclinepi.2020.05.001. Epub 2020 May 11. PMID 32438024